CLINICAL TRIAL: NCT03156348
Title: Impact of Clinical Pharmacist on Post-discharge Prevention of Adverse Drug Events in Older Adults: Randomized Clinical Trial.
Brief Title: Impact of Clinical Pharmacist on Adverse Drug Events in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Marcela Jirón Aliste, associate proffesor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SA14ID0141
Record Dates: First submitted 2017-05-10; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Drug-Related Side Effects and Adverse Reactions
Keywords: Pharmaceutical intervention; Older adult; Internal medicine; Adverse drug event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: parallels groups: control arm will receive usual care, intervention arm will receive a Clinical Pharmacist Care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervented (Experimental): The intervention group will receive in addition to the usual care, it will receive the Clinical Pharmacist Care during hospitalization, discharge and during 2 months post-discharge, through a home visit at 30 ± 5 days post-discharge and a telephone call at 60 ± 5 days.
  Interventions: Other: Clinical Pharmacist Care
- Control (No Intervention): The control group will receive hospital care and discharge from a clinical team previously trained in geriatric clinical pharmacology, which includes epicrisis, indications that the physician deems pertinent to the discharge and prescriptions if necessary and a medical control at 15 days post-discharge.
  Information will be collected that allows the characterization:
  * Sociodemographic
  * Morbid
  * Pharmaco-therapeutic
  * Functionality before (baseline), during and after hospitalization
  A physician, a pharmacist and an occupational therapist, blind to the treatment assignment, will collect the records using a specially designed record. Post-discharge evaluations will be conducted through telephone interviews at 30, 60 and 90 days after hospital discharge.

INTERVENTIONS:
Other: Clinical Pharmacist Care — During hospitalization and at discharge a clinical pharmacist (CP) will monitor daily pharmacological safety and efficacy of the medication to asses and make appropriate recommendations. CP will explain the use reasons of each of the drugs.
  At 30 days post-discharge, the CP will review the updated clinical record of patient and conduct a home visit to enhance and ask about adherence, self-medication, medication use at that time and possible results of laboratory tests performed and clarify doubts regarding the use of current medications. The same activities will be made at 60 days by telephonic way, to reinforce the recommendations.
  Arms: Intervented

SUMMARY:
Adverse drug events (ADE) are one of the major problems affecting quality of care and achievement of therapeutic goals in older adults (OA), increasing re-admissions, hospital stays, resource use, and problems on patient safety. The present study aim is to determine the impact of the clinical pharmacist interventions on the prevention of ADE in OA at 3 months post-discharge compared to usual care.

A randomized clinical trial of two parallel groups 1: 1 (control and intervention) plus a historical control group will be carried out at the Internal Medicine Service (IMS) of the teaching Hospital at the University of Chile. The sample will be of 611 patients (242 per each parallel group and 127 of the historical control group) of 60 years or older, admitted to the IMS for acute pathology or decompensation of chronic pathology, with survival over 6 months, who is under pharmacological therapy and have a caretaker or responsible contact person at discharge.

The historical control group will receive usual care and the parallel control group will also receive training on pharmacogeriatrics. The intervention group will receive the care of a clinical pharmacist during hospitalization, at discharge and post-discharge, through a home visit at 30 days post-discharge and a telephone call at 60 days post discharge.

DETAILED DESCRIPTION:
The intervention plan during hospitalization will consist of daily monitoring of pharmacological efficacy and safety, participating in clinical rounds and patient interviews. To review, assess the indications according to the conditions of each patient and evaluating possible interactions of clinical importance, dose adjustments, potentially inappropriate medication for older adult (OA), adverse effects and omissions of therapy. To make recommendations to the healthcare team regarding pharmacological therapy received during hospitalization and at discharge.

Patient-directed interventions will occur at discharge and post-discharge, focusing on clarifying management regimens, drug use motives, preventing drug-related problems, clarifying doubts and educating on pharmacotherapy, and enhancing adherence to treatment. The selection and recruitment of the patients will be made during the first 48 hours of their admission to the Internal Medicine Service (IMS), where they will be invited to participate and sign the informed consent.

In all groups, a physician, pharmacist, and occupational therapist, blind to treatment assignment, will collect sociodemographic, morbid, pharmacotherapeutic, and functional (Barthel Index and Lawton & Brody Scale), adherence (Morisky & Green Scale), delirium (Confusion Assessment Method, CAM), comorbidity (cumulative illness rating scale in Geriatrics (CIRS-G)), anticholinergic burden (Anticholinergic Burden Scale and Ars Risk Scale), potentially inappropriate medications (Beers Criteria and screening tool of older people's prescriptions & screening tool to alert to right treatment criteria (STOPP & START)) before, during hospitalization, at discharge and post-discharge. Also a follow up by telephone interviews at 30, 60 and 90 days after hospital discharge from the IMS.

Two trained and independent evaluators (geriatrician and clinical pharmacist), blind to treatment assignment, will evaluate the history of each case and by consensus will assign the presence of Adverse Drug Events (ADE), and classify them as preventable or not and according to severity. The Chi-squared or Fisher exact test will be used to test the hypothesis that clinical pharmacist intervention prevents at least 50% of ADE at 3 months post-discharge in OA compared to usual care in the IMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients attended by the staff of internists of the internal medicine service of the Clinical Hospital of the University of Chile for acute condition or decompensation of chronic pathology.
* Patients with an estimated survival of more than 6 months.
* Patients who are on pharmacological therapy.
* Patients who have a contact person or responsible caregiver, willing to comply with the scheduled care plan.
* Patients who have a contact telephone number

Exclusion Criteria:

* Patients without cognitive autonomy in which it is not possible to establish contact with the caregiver.
* Any other condition that in the judgment of the research team affects the quality of the collection of the information.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Estimated)
Dates: Start 2015-05-02 (Actual); Primary Completion 2017-09-22 (Estimated); Study Completion 2017-12-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Drug Events at 90 days post discharge | 90 days post discharge
  Two trained and independent evaluators (geriatrician and clinical pharmacist), blind to treatment allocation, will evaluate the history of each case and by consensus will assign the presence of ADE, and classify them as preventable or not preventable and according to severity.

SECONDARY OUTCOMES:
Adherence measured with Morisky & Green Scale | 90 days post discharge
  test with 4 question to know adherence to treatment of the patient
Incidence of potentially inappropriate medication | 90 days post discharge
  The evaluation of which drugs will be considered inappropriate will be performed according to the Beers criteria and STOPP & START criteria, both allow to evaluate if the indicated medicines are appropriate for the older adults.
Incidence of adverse drug reactions | 90 days post discharge
  The analysis of the direct relationship between adverse reaction and drug use, will be determined by a multidisciplinary team following validated instruments.
Incidence of non-programmed/programmed consultations or hospitalizations after discharge from the hospital | 90 days post discharge
Prevalence of Polypharmacy (5 or more drugs) | 90 days post discharge
  polypharmacy is a risk factor for many clinical outcomes related with treatment failure or drug related problems
Prevalence of self medication in each group | 90 days post discharge
  when patient take a drug without medical indications, it is considerate self medication.
Presence of clinically relevant drug interactions | 90 days post discharge
  Clinical relevance will be discussed with a multidisciplinary group
Characterization of the interventions made by the clinical pharmacist to the health team | 90 days post discharge
  Cinical phasrmacist interventions may be:
  * Dose adjustments
  * Change, addition or withdrawal of a drug
  * change in treatment regimen or schedule
  * Medication errors prevention
  * Drug-drug Interactions prevention
  * Patient or health team education.
  * Actions to improve the clinical outcome of the patients.
  Interventions relevance will be discussed with a multidisciplinary group

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Jirón, PhD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico de la Universidad de Chile, Independencia, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No